CLINICAL TRIAL: NCT00319267
Title: An Open Label, Multicenter Study to Assess the Pharmacokinetics, Tolerability, and Safety of a Pediatric Formulation of Bosentan in Children With Idiopathic or Familial Pulmonary Arterial Hypertension
Brief Title: Bosentan in Children With Pulmonary Arterial Hypertension
Acronym: FUTURE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-365; 2004-005157-63 (EudraCT Number)
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: bosentan; children; pharmacokinetics; pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan

ARMS (1):
- Bosentan (Experimental): The initial dose of bosentan was 2 mg/kg b.i.d. for 4 weeks. After 4 weeks, the initial dose was up-titrated to the maintenance dose of 4 mg/kg b.i.d. up to the end of the study treatment at Week 12. If the maintenance dose was not well tolerated, the dose could be down-titrated to the initial dose.
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — Pediatric oral formulation of bosentan, i.e., 32 mg dispersible and breakable tablets
  Other Names: ACT-050088; Ro 47-0203

SUMMARY:
The aim of the study is to demonstrate that the exposure to bosentan in children with idiopathic pulmonary arterial hypertension (PAH) or familial pulmonary arterial hypertension, using a pediatric formulation, is similar to that in adults with PAH and to evaluate the tolerability and safety of a pediatric formulation of bosentan in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the parents or the legal representatives.
* Males or females >= 2 and < 12 years of age.
* Idiopathic PAH or familial PAH diagnosed by right heart catheterization (Clinical classification of pulmonary hypertension, Venice 2003).
* World Health Organization (WHO) functional class II or III.
* Oxygen saturation (SpO2) >= 88% (at rest, on room air).
* PAH treatment-naïve patients or patients already treated with either:

  * Bosentan monotherapy
  * Intravenous epoprostenol monotherapy
  * Intravenous or inhaled iloprost monotherapy
  * Combination of bosentan and intravenous epoprostenol
  * Combination of bosentan and intravenous or inhaled iloprost.
* All patients should start the study drug (bosentan pediatric formulation) at 2 mg/kg twice daily (b.i.d.), whether or not they were previously treated with bosentan.
* PAH therapy stable for at least 3 months prior to Screening.
* Stable treatment with calcium channel blockers, if any, for at least 3 months prior to Screening.
* Patient's PAH condition stable for at least 3 months prior to Screening.

Exclusion Criteria:

* PAH associated with conditions other than idiopathic or familial PAH.
* Non-stable patients, e.g., history (in the last 3 months prior to Screening) of recurrent syncope, or signs and symptoms of non-compensated right heart failure.
* Need or plan to wean patients from intravenous epoprostenol, or intravenous, or inhaled iloprost.
* Body weight < 4 kg.
* Systolic blood pressure < 80%, the lower limit of normal range, according to age and gender.
* AST and/or ALT values > 3 times the upper limit of normal ranges.
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.
* Hemoglobin and/or hematocrit levels < 75% of the lower limit of normal ranges.
* Pregnancy.
* Known intolerance or hypersensitivity to bosentan or any of the excipients.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2005-05; Primary Completion 2006-12 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve during a dose interval (AUCt) for bosentan | At pre-dose and 0.5h, 1h, 3h, 7.5h, and 12h post-dose
  AUCt was assessed at steady state (i.e., after at least 2 weeks of treatment with a same dose of the study drug) over 12 hours .

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of bosentan and its metabolites | At pre-dose and 0.5h, 1h, 3h, 7.5h, and 12h post-dose
  Maximum observed plasma concentration for bosentan and its metabolites was directly derived from their respective plasma concentration-time curves.
Time to reach the maximum plasma concentration (tmax) of bosentan and its metabolites | At pre-dose and 0.5h, 1h, 3h, 7.5h, and 12h post-dose
Area under the plasma concentration-time curve during a dose interval (AUCt) for the metabolites of bosentan | At pre-dose and 0.5h, 1h, 3h, 7.5h, and 12h post-dose
  AUCt was assessed at steady state (i.e., after at least 2 weeks of treatment with a same dose of the study drug) over 12 hours.

REFERENCES:
- [Result] Beghetti M, Haworth SG, Bonnet D, Barst RJ, Acar P, Fraisse A, Ivy DD, Jais X, Schulze-Neick I, Galie N, Morganti A, Dingemanse J, Kusic-Pajic A, Berger RM. Pharmacokinetic and clinical profile of a novel formulation of bosentan in children with pulmonary arterial hypertension: the FUTURE-1 study. Br J Clin Pharmacol. 2009 Dec;68(6):948-55. doi: 10.1111/j.1365-2125.2009.03532.x. PMID 20002090